CLINICAL TRIAL: NCT01759836
Title: A Randomized Double Blind, Placebo-controlled Study Determining the Role of Adjuvant Statin Therapy in Patients Who Underwent Radical Prostatectomy for Locally Advanced Prostate Cancer
Brief Title: Impact of Adjuvant Statin Therapy in Patients Who Underwent Radical Prostatectomy for Locally Advanced Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Dong-A Pharmaceutical (Industry)
Responsible Party: Principal Investigator, In Gab Jeong, MD, professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AMC-PC2012002
Record Dates: First submitted 2013-01-01; First posted 2013-01-03 (Estimated); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Prostatic Neoplasms
Keywords: Prostatectomy; Statins
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atorvastatin 20mg (Experimental): Atorvastatin 20mg daily for 1 year
  Interventions: Drug: Atorvastatin 20mg
- Placebo (Placebo Comparator): Placebo daily for 1 year
  Interventions: Drug: Atorvastatin 20mg

INTERVENTIONS:
Drug: Atorvastatin 20mg — Atorvastatin 20mg daily for 1 year

SUMMARY:
Biochemical recurrence develops in approximately 30-40% of men with locally advanced prostate cancer who undergo radical prostatectomy. To date, the effect of statins on prostate cancer recurrence has been investigated in several retrospective studies with inconsistent results. The purpose of this study is to determine the impact of statin on biochemical recurrence after radical prostatectomy for locally advanced prostate cancer.

DETAILED DESCRIPTION:
Estimated Enrollment: 354

Study start date: October 2012

Estimated Study Completion Date: October 2015

Statin Group: Treatment with Atorvastatin 20mg daily after radical prostatectomy during 1 year.

Control Group: Treatment with Placebo daily after radical prostatectomy during 1 year.

Follow up: every 3 months for the first year. Check PSA, Total/LDL-cholesterol and Triglyceride.

Primary End Point Rate of Biochemical recurrence

Secondary End Point Clinical progression of prostate cancer Change of Total/LDL- cholesterol and Triglycerides 5 year-Biochemical recurrence free survival

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have correspond to one of the following three pathologic criteria.

   A. Gleason scores 8 or greater B. Positive resection margin C. pT3-T4
2. Patients must have pathologically adenocarcinoma
3. Patients must be enrolled within 60 days after radical prostatectomy
4. Patients must be able to provide written informed consent

Exclusion Criteria:

1. Patients who have received neoadjuvant androgen deprivation therapy
2. Patients who have the participation of other clinical trial within the past 3 months
3. Patients who have treated with statin
4. Patients who have lymph node metastasis or distant metastasis
5. Patients who have 10 year risk of cardiovascular disease over 10% based on NCEP ATP III guideline.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 364 (Actual)
Dates: Start 2012-10; Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Rate of biochemical recurrence | One year

SECONDARY OUTCOMES:
Biochemical recurrence free survival | Five years

OTHER OUTCOMES:
Clinical progression-free survival | Five years

CONTACTS AND LOCATIONS:
Overall Officials: Choung-Soo Kim, MD, Principal Investigator — Department of Urology,Asan Medical Center, Seoul
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Background] Jeong IG, Lim B, Yun SC, Lim JH, Hong JH, Kim CS. Adjuvant Low-dose Statin Use after Radical Prostatectomy: The PRO-STAT Randomized Clinical Trial. Clin Cancer Res. 2021 Sep 15;27(18):5004-5011. doi: 10.1158/1078-0432.CCR-21-0480. Epub 2021 May 19. PMID 34011557